CLINICAL TRIAL: NCT05400200
Title: Study of the Involvement of Cognitive, Emotional, and Behavioural Self-regulation and Control Capacities in the Modulation of Post-traumatic Stress Disorder Symptomatology in Adults: Processual and Integrative Approach
Brief Title: PTSD and Self-regulation: Coping, Emotional Regulation and Cognitive Control and Their Relationships to Symptom Management
Acronym: RESIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-PP-29
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: post-traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- questionnary with patients Definite diagnosis of PTSD (Other): only patients with diagnosis of PTSD answered questionaries
  Interventions: Diagnostic Test: questionnary administration

INTERVENTIONS:
Diagnostic Test: questionnary administration — questionary

SUMMARY:
Non-pathological stress has an adaptive value, allowing a person to prepare for the demands of everyday life and increasing chances of survival in the face of danger. To "cope", the individual responds with behavioural, emotional and cognitive strategies (coping strategies). Coping aims to modify the problem causing the stress (problem-focused coping) or to regulate the emotional responses associated with the problem (emotion-focused coping), or it can be focused on avoidance (psychologically and/or physically avoiding the source of the stress). Coping is therefore not positive or negative per se and the strategies used by an individual can be positively or negatively associated with resilience. Thus, the mechanisms by which coping strategies, whether dispositional or situational, induce resilience or, conversely, the development of symptoms linked to stress and PTSD remain poorly understood.

To detect and characterize some of these mechanisms, the present research focuses on high-level capacities closely linked to coping and resilience and involved in stress and psychotrauma, namely cognitive control (notably attentional and executive processes that allow for adaptive control of cognition and behaviour) and emotional regulation (processes allowing the triggering, inhibition, maintenance or modulation of emotions). The global research program includes different studies aimed at analyzing and screening for factors, or complexes of factors, that may be involved in the modulation of PTSD symptomatology in adults, based on a dimensional process-oriented and integrative approach. The present study will examine the relationship between the severity and nature of the symptoms of PTSD (e.g. avoidance) and the different processes considered. The primary objective is to examine the impact of the preferential use of habitual coping strategies (emotion-focused, problem-focused or avoidance-focused coping) on the severity of PTSD symptoms. Another objective is to explore the interrelationships, in the modulation of symptoms, between these (specific) coping strategies and the more general and stable self-regulatory capacities, namely emotional regulation and cognitive control. 50 patients aged between 18 and 65 years, followed for a definite diagnosis of PTSD, will participate and complete a set of self-questionnaires and neuropsychological tests.

DETAILED DESCRIPTION:
Numerous epidemiological studies confirm that psychological trauma is a ubiquitous phenomenon and many researchers consider exposure to trauma to be the norm rather than the exception. However, not all individuals exposed to a traumatic event will develop PTSD and not all will react in the same way to an identical event: some may be resilient while others will develop symptoms of varying nature, intensity and duration.

PTSD symptoms are often seen as a stress response that remains disrupted and maladaptive in the absence of the event that provoked it, and some approaches view reactions to psychotrauma along a continuum from a normal coping response to stress to chronic PTSD.

Non-pathological stress has an adaptive value, allowing a person to prepare for the demands of everyday life and increasing the chances of survival in the face of danger. To "cope", the individual responds with behavioural, emotional and cognitive strategies (coping strategies). Conceived as a moderator of the stressful event/emotional distress relationship, coping is defined by classical approaches as a multidimensional, dynamic and specific process and not a general and stable characteristic.

Recently, a second way of modelling coping has emerged, which refers to dispositional adjustment (or trait adjustment) and assumes that individuals develop habits for coping with stress and threat and that these habits or adjustment styles can affect their response in new situations. The latter approach seems to be more appropriate because dispositional coping measures are shown to be more stable over time.

Coping can be used to modify the problem causing the stress (problem-focused coping) or to regulate the emotional responses associated with the problem (emotion-focused coping), or it can be focused on avoidance (psychologically and/or physically avoiding the source of the stress). It is therefore not positive or negative per se, and the strategies used by an individual can be positively or negatively associated with resilience. To date, however, the mechanisms by which coping strategies, whether dispositional or situational, induce resilience or, conversely, the development of symptoms linked to stress and PTSD remain poorly understood.

Firstly, emotions are inherent to stress and trauma and their regulation is initiated to reduce an unpleasant experience in order to produce an adapted behaviour. In addition, cognitive control is involved whenever we have to deal with new and/or complex situations that we cannot solve automatically and routinely, which is the case when confronted with a traumatic event. It is thus clear that emotional regulation and cognitive control must be efficient to deal with such exceptional events as traumatic ones.

In order to detect and characterize some of these mechanisms, the present research project focuses on high-level capacities closely linked to coping and resilience and involved in stress and psychotrauma, namely cognitive control and emotional regulation.

The main study examines the impact of the preferred use of habitual coping strategies (emotion-focused, problem-focused or avoidance-focused coping) on the severity of PTSD symptoms. The secondary objective is to explore the interrelationships, in the modulation of symptoms, between these (specific) coping strategies and the more general and stable self-regulatory capacities, namely emotional regulation (processes allowing the triggering, inhibition, maintenance or modulation of emotions) and cognitive control (notably attentional and executive processes that allow for adaptive control of cognition and behavior). The study will examine the relationship between the severity and nature of the symptoms of PTSD (e.g. avoidance) and the different processes considered. Fifty patients aged between 18 and 65 years, followed for a definite diagnosis of PTSD, will participate in this study and will complete a set of self-questionnaires and neuropsychological tests.

Despite their importance, and despite the many characteristics that cognitive control, emotional regulation and coping may share, research on these concepts has remained particularly fragmented, not studying these three essential facets together. In an original way, the approach adopted in this project is processual and integrative and considers a set of processes underlying these capacities. A better understanding of these influences on vulnerability to psychological trauma may help to refine conceptual models of PTSD, as each of these factors considered in isolation is likely to play only a small role in the overall resilience capacity or risk of PTSD. A more integrative consideration of stress and trauma management factors may thus help to improve the management and early identification of risk for adverse clinical outcomes and thus alert clinicians to those who may be most in need of prevention or early intervention following exposure to an extremely stressful and/or traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of PTSD
* Aged between 18 and 65
* Stable medication for at least 2 weeks
* Understand, speak and read French fluently
* Having signed the informed consent form
* Being affiliated to the social security system

Exclusion Criteria:

* Medical condition that would interfere with the ability to give consent and participate in the study
* Presence of a mental condition with suicidal risk that requires priority treatment or care
* Severe psychiatric comorbidity: schizophrenia; bipolar disorder; severe depression
* Neurological disorders
* Intellectual disability
* Pervasive developmental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
PTSD severity score : total score of the PCL-5 (Posttraumatic stress disorder Checklist). | Day 0
  20-item self-report questionnaire that assesses the presence and intensity of PTSD symptoms according to DSM-5 criteria and provides an overall PTSD severity score

SECONDARY OUTCOMES:
PTSD clusters' severity scores | day 0
  total score of each sub-scale of the PCL-5.

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL BENOIT, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France, France

IPD SHARING:
Plan to Share IPD: No